CLINICAL TRIAL: NCT06942364
Title: The Effect of Action Observation Therapy on Balance and Lower Extremity Function in Children With Hemiparetic Cerebral Palsy
Brief Title: Action Observation Therapy in Hemiparetic CP: Impact on Balance & Lower Limb Function
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fatih Tekin (Other)
Responsible Party: Sponsor-Investigator, Fatih Tekin, Assist. Prof., Pamukkale University
Organization: Pamukkale University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Action Observation Therapy
Record Dates: First submitted 2025-04-10; First posted 2025-04-24 (Actual); Last update posted 2025-04-24 (Actual); Status verified 2025-04

CONDITIONS: Hemiparetic Cerebral Palsy Children
Keywords: Action Observation Therapy; Hemiparetic Cerebral Palsy; Balance; Lower Extremity Function; Rehabilitation

STUDY DESIGN:
Intervention Model Description: The discovery of the mirror neuron system's role in motor learning has led to the development of Action Observation Therapy (AOT). In AOT, patients observe a video of specific movements or watch an instructor perform actions, then attempt to imitate them. This rehabilitation strategy is designed to repair damaged neural networks and re-establish motor function in individuals with central nervous system lesions. While several studies have shown that AOT can improve upper extremity function and reaching performance in children with CP, there is limited evidence regarding its effects on lower extremity function. Notably, no studies from our country have investigated the impact of AOT on balance and lower extremity function in children with CP.
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- experimental (Experimental)
  Interventions: Other: Action Observation Therapy; Other: conventional physiotherapy
- control (Active Comparator)
  Interventions: Other: conventional physiotherapy

INTERVENTIONS:
Other: Action Observation Therapy — The AOT video comprised four specific tasks designed to improve lower extremity function, balance, and gait (Figure 1):
  1. Sitting Balance: Movements to enhance balance while seated (Figure 2).
  2. Sit-to-Stand Transition: Exercises to facilitate the transition from sitting to standing.
  3. Walking and Balance: Gait and balance training on a parallel bar or flat surface.
  4. Single-Leg Balance: Activities focused on improving balance on one leg. For each task, children observed the movement for 1 minute, then practiced the action for 5 minutes. A 1-minute rest period was allowed between tasks, with a total AOT session lasting 30 minutes. All sessions were conducted by the same physiotherapist.
  Arms: experimental
Other: conventional physiotherapy — Conventional physiotherapy is a widely used therapeutic approach that focuses on improving physical function, mobility, and overall quality of life through evidence-based techniques. It typically includes exercises for strength, flexibility, balance, and coordination, along with manual therapy, postural training, and education about movement and body mechanics. This traditional method is commonly applied in the rehabilitation of patients with neurological, orthopedic, and musculoskeletal conditions. In pediatric populations, such as children with cerebral palsy, conventional physiotherapy plays a vital role in promoting motor development, enhancing functional independence, and preventing secondary complications.

SUMMARY:
Background:

Action Observation Therapy (AOT) leverages the mirror neuron system to enhance motor learning and is anticipated to improve upper extremity function in children with cerebral palsy. However, its effects on balance, lower extremity function, and gait performance in children with hemiparetic cerebral palsy remain underexplored. The planned study aims to evaluate whether the addition of AOT to conventional physiotherapy will positively influence balance, lower extremity function, and gait performance in this population.

Objective:

The study is designed to assess the efficacy of incorporating AOT as an adjunct to conventional physiotherapy in improving balance, lower extremity function, and gait performance in children with hemiparetic cerebral palsy.

Methods:

A patient cohort consisting of children with hemiparetic cerebral palsy (GMFCS levels I and II) is planned to be assembled.

It is expected that a total of 20 patients will be recruited and then randomly allocated into an experimental group and a control group.

The experimental group is scheduled to receive conventional physiotherapy in addition to AOT sessions, while the control group is planned to receive conventional physiotherapy only.

The intervention period is planned for 6 weeks, during which both groups will participate in 12 physiotherapy sessions.

Additionally, the experimental group is scheduled to undergo AOT sessions twice weekly, with each session lasting 30 minutes.

Outcome measures to be employed will include the Timed Up and Go (TUG) test, Pediatric Balance Scale, Five-Step Stair Climbing and Descending Test, and the 6-Minute Walk Test (6MWT).

This study is expected to systematically evaluate the potential benefits of adding AOT to standard physiotherapy regimens for enhancing balance, lower extremity function, and gait performance in children with hemiparetic cerebral palsy.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed hemiparetic type of cerebral palsy

Exclusion Criteria:

* Any other types of cerebral palsy

Ages: 5 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 20 (Actual)
Dates: Start 2023-01-10 (Actual); Primary Completion 2024-06-10 (Actual); Study Completion 2024-12-10 (Actual)

PRIMARY OUTCOMES:
Timed Up and Go Test | This test will be administered twice: once before and once after a 6-week intervention period comprising a total of 12 sessions.
  The Timed Up and Go (TUG) Test is a simple and widely used clinical tool to assess a person's mobility, balance, and risk of falling. It involves timing a person as they rise from a standard chair, walk a distance of 3 meters, turn around, walk back to the chair, and sit down. The total time taken to complete this sequence is recorded, with shorter times generally indicating better functional mobility. The TUG Test is commonly used in various populations, including older adults and individuals with neurological conditions such as stroke or cerebral palsy, to evaluate progress during rehabilitation or to identify individuals at risk of falls. It is valued for its ease of use, minimal equipment requirements, and ability to reflect real-world functional movements.
Pediatric Balance Scale | This test will be administered twice: once before and once after a 6-week intervention period comprising a total of 12 sessions.
  A modified version of the Berg Balance Scale for children, the PBS consists of 14 items (maximum score 56). It assesses functional balance through activities such as sitting-to-standing, standing, transfers, stepping, single-leg stance, turning, bending, and reaching. The scale has demonstrated strong correlations with other functional measures in children with CP
Five-Step Stair Climbing and Descending Test | This test will be administered twice: once before and once after a 6-week intervention period comprising a total of 12 sessions.
  This test evaluates functional mobility parameters including walking speed, strength, active joint range, and balance. Children are instructed to ascend and descend a 5-step staircase without pausing. The better of two trials is recorded; a shorter completion time indicates superior functional performance
6-Minute Walk Test | This test will be administered twice: once before and once after a 6-week intervention period comprising a total of 12 sessions.
  Originally developed by Balke (1963), the 6MWT measures the distance walked in 6 minutes, reflecting the child's functional capacity for daily activities. In children with CP, typical distances range from 334 to 455 meters, varying according to sex, age, height, weight, and step length

CONTACTS AND LOCATIONS:
Locations (1):
- Pamukkale University Faculty of Physiotherapy and Rehabilitation, Denizli, Kınıklı, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No